CLINICAL TRIAL: NCT06359457
Title: Correlation Between Serum Progesterone Level And Menstrual Symptoms In Young Females With Primary Dysmenorrhea
Brief Title: Correlation Between Serum Progesterone Level And Primary Dysmenorrhea
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennaallah Yousef Mohamed Nasreldien, Lecturer of physical therapy for women's health, Cairo University
Other Study IDs: P.T.REC/012/005016
Record Dates: First submitted 2024-03-30; First posted 2024-04-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-04

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhoea; Serum progesterone level; Visual analogue scale; Menstrual symptoms questionnaire
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A group of young females with primary dysmenorrhea: One hundred young females with primary dysmenorrhea will participate in this study. They will be recruited from the Gynecological outpatient clinic, Kasr El Ainy University Hospital, Cairo, Egypt.
  All females should have regular menstrual cycles. Taking blood samples of 3 ml through the cubital vein to examine the levels of serum progesterone will be carried out on the 21st day of menstruation, while to assess the pain intensity of primary dysmenorrhea using the Visual Analogue Scale (VAS) and physical and psychological symptoms associated with dysmenorrhea will be assessed by menstrual symptoms questionnaire
  .

SUMMARY:
This study will be conducted to determine the correlation between the levels of serum progesterone and Menstrual Symptoms In Young Females with primary dysmenorrhea.

DETAILED DESCRIPTION:
One hundred adult females with primary dysmenorrhea will participate in this study. They will be recruited from the Gynaecological outpatient clinic, Kasr El Ainy University Hospital, Cairo, Egypt Many studies reported that primary dysmenorrhea was the result of increased prostaglandin, especially prostaglandin F2α (PGF2α) and prostaglandin E2 (PGE2) which produced the effect through the cyclooxygenase pathway, and further led to uterine ischemia hypoxia. Nevertheless the relationship between the serum progesterone level and menstrual symptoms was not completely clear. Hence, this study will investigate the association between the serum progesterone level and menstrual symptoms in young females with primaryf dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

1. One hundreds adult females were suffered from primary dysmenorrhea.
2. Their age was ranged from 17 to 24 years.
3. Their body mass index was ranged from 20 to 25 kg/m2.

Exclusion Criteria:

* Any participant will be excluded from the study if they have:

  1. Irregulars or infrequent menstrual cycles.
  2. Pacemaker, Myasthenia gravis, hyperthyroidism, active tuberculosis and psychosis.
  3. Pelvic pathology.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: One hundred girls with dysmenorrhoea. Menarche at least 3 years ago. All females should be regular menstrual cycles.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Serum progesterone level | 1 month
  Blood samples will be taken by physician for each girl, and will send to laboratory center to measure the progesterone level in the blood. The normal serum progesterone level at 21st day is 4-20 ng
Pain intensity | 1 month
  It will be measured by Visual analogue scale. It is 10 cm line with values ranging from 0 to 10. 0 indicates no pain nd 10 indicates the worst pain.
Physical and psychological menstrual symptoms | 1 month
  It will be measured by menstrual symptoms questionnaire. It is 25 items split into two categories which used to assess the physical and psychological symptoms associated with dysmenorrhea. The score on each item ranged from 1 (never) to 5 (always) with a higher composite score indicating more symptoms
Correlation between serum progesterone level and pain | 1 month
  The correlation between serum progesterone level and pain intensity measured by the VAS will be conducted
Correlation between serum progesterone level and menstrual symptoms | 1 month
  The correlation between serum progesterone level and menstrual symptoms measured by the menstrual symptom questionnaire will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: HANAA HAFEZ, PhD, Study Director — Lecturer of Physical Therapy for Orthopedic. Physical Therapy, Nahda University.; RANIA Hamed, PhD, Study Director — Lecturer of Physical Therapy for Basic Science. Physical Therapy, Nahda University.; ESRAA MOHAMED, PhD, Study Director — Lecturer Of Physical Therapy For Cardiovascular, Respiratory and Geriatrics.; HOSSAM HUSSIEN, PhD, Study Director — Faculty of Medicine, Al-Azhar University.
Locations (1):
- Menna Allah Youssef Nasr El-Dien, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided